CLINICAL TRIAL: NCT04527159
Title: Comparison Between Two Different Desensitizing Materials in Controlling Natural Dentin Hypersensitivity: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Desensitizing Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourah Mulfi Aljasser (Other)
Responsible Party: Sponsor-Investigator, Nourah Mulfi Aljasser, Principal Investigator, Riyadh Elm University
Organization: Riyadh Elm University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: dentin hypersensitivity
Record Dates: First submitted 2020-08-19; First posted 2020-08-26 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — VivaSens Liner

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- desensitizing agents (Fluoraphat Pro and VivaSens®) (Other): 22 participants above the age of 18 years who presented to dental clinics in Riyadh Elm University with dentine hypersensitivity were randomly selected to participate in the study.
  Each participant has at least two teeth with natural hypersensitivity which was not caused by any iatrogenic causes or bad oral habits, so there are 44 cases divided into two groups according to the material used, each group has 22 teeth, that make it applicable to apply the studied material with every patient on individual tooth with the same variables of the oral mouth. When teeth in the hypersensitivity group were evaluated for the level of DH, all teeth were found to have Grade 4 sensitivity.
  Interventions: Drug: Fluoraphat Pro / VivaSens

INTERVENTIONS:
Drug: Fluoraphat Pro / VivaSens — desensitizing agents for treatment of dentinal hypersensitivity
  Other Names: VivaSens

SUMMARY:
To compare the efficacy of two commercially available in-office desensitizing agents (Fluoraphat Pro and VivaSens®), in the treatment of dentinal hypersensitivity.

DETAILED DESCRIPTION:
Dentine hypersensitivity (DH) is a condition that occurs in non-pathological, non-defective teeth and is defined as "a short, sharp pain in response to stimuli, typically thermal, evaporative, tactile, osmotic or chemical and which cannot be attributed to any other dental defect or pathology". The incidence of DH ranges from 4% to 74% in several studies. Mandibular first molars, canines and premolars of both jaws are most commonly affected by DH.

The pathogenesis of DH is linked to exposure of dentinal tubules that can occur in the oral cavity due to dental erosion from acidogenic diets, aggressive tooth-brushing, injudicious use of whitening products, gingival recession, periodontal debridement or surgery. The most commonly reported initiating factor is cold drinks. Management usually involves methods that can achieve one or both of the following objectives; i) alteration of fluid flow in the dentinal tubules and ii) modification or blocking of the pulpal nerve response.

A broad range of products that achieve these objectives have been developed after rigorous trials and can be used in-office or at home depending on the severity of the condition. These products are commonly referred to as desensitizing agents. Grossman suggested that an ideal desensitizing agent should be non-irritating to the pulp, relatively painless on application, easy to apply, rapid in action, effective for long periods of time and should not stain the teeth.

The use of dentine desensitizers has become one of the most common methods in managing DH. The most commonly used desensitizers contain components such as fluoride, triclosan, benzalkonium chloride, ethylene diaminetetraacetic acid and glutaraldehyde. Fluoraphat Pro (Neumunster, Germany) and VivaSens® (Ivoclar Vivadent, Schaan, Liechtenstein, Switzerland) are two agents that have been tested for use as dentine desensitizers and are currently available for commercial use. In the present study, two such varnishes VivaSens (Ivoclar Vivadent, Schaan, Liechtenstein, and Switzerland) and Fluoraphat (Promedical Neumunster, Germany) have been used. The present study aims to establish which of the two desensitizing agents has better efficacy in reducing hypersensitivity in patients who have been previously diagnosed with DH.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 50 years
* Patient should have at least 2 teeth with dentinal hypersensitivity
* Sound tooth structure
* Willingness to participate in the study

Exclusion Criteria:

* Gingival recession
* Caries
* Non-carious lesions (attrition, abrasion, erosion, abfraction)
* Teeth restored with dental filling
* Fractured or cracked tooth
* Microleakage

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender and Age are not included in the calculation, since the effects could not be determined reliably
Enrollment: 22 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Likert type scale used to measure attitudes or opinions | 24 Hours
  Likert type scale grading from 0-4 0: No sensitivity
  1. Very mild sensitivity
  2. Mild sensitivity
  3. Moderate Sensitivity
  4. Severe Sensitivity to compare the efficacy of two commercially available in-office desensitizing agents (Fluoraphat Pro and VivaSens®), in the treatment of dentinal hypersensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Roula Alboouni, Prof, Study Director — Riyadh Elm University
Locations (1):
- Nourah Aljasser, Riyadh, Saudi Arabia